CLINICAL TRIAL: NCT00012168
Title: Lymphoscintigraphy Assisted Molecular Staging of Head and Neck Cancer
Brief Title: Lymphoscintigraphy to Detect Early Metastases in Patients With Cancer of the Mouth or Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000068489; NYU-9917; NCI-G01-1915
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: stage 0 oropharyngeal cancer; stage 0 lip and oral cavity cancer; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — iso-sulfan blue; Polymerase Chain Reaction; Immunohistochemistry; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

INTERVENTIONS:
Drug: isosulfan blue
Genetic: polymerase chain reaction
Other: immunohistochemistry staining method
Procedure: lymphangiography
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: New imaging procedures such as lymphoscintigraphy may improve the ability to detect the spread of mouth and throat cancer to lymph nodes in the neck.

PURPOSE: Pilot study of lymphoscintigraphy followed by sentinel lymph node mapping and sentinel lymph node biopsy to detect lymph node metastases in the neck in patients who have mouth or throat cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the sensitivity of lymphoscintigraphy and isosulfan blue in localization of sentinel lymph nodes in patients with previously untreated squamous cell carcinoma of the oral cavity or oropharynx.
* Determine evidence of micrometastases in histologically normal sentinel lymph nodes resected from these patients.
* Assess the clinical significance of micrometastases in lymph nodes resected from these patients.

OUTLINE: Patients undergo preoperative lymphoscintigraphy utilizing technetium Tc 99m sulfur colloid followed by intraoperative injections of isosulfan blue at 3-4 locations into the primary tumor periphery. Once the afferent lymphatic channel and sentinel node have been identified, patients undergo cervical lymphadenectomy followed by resection of the primary tumor.

Resected primary tumor, radioactive lymph nodes, and blue-stained sentinel nodes are then subjected to molecular (polymerase chain reaction) and histocytochemical (immunohistochemistry for cytokeratin and micrometastases, light microscopy) analyses.

Patients are followed at 1, 3, 6, 12, 18, and 24 months.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary squamous cell carcinoma of the oral cavity or oropharynx

  * Stage 0-IVA (Any T, N0)
* No low-risk tumors
* Must require elective staging neck dissection and resection of primary tumor

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No concurrent impaired mental status

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No prior surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moni A. Kuriakose, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States